CLINICAL TRIAL: NCT05342805
Title: Comparison of Subtotal Stomach and Narrow Gastric Tube for Reconstruction After Esophagectomy for Gastric Cancer: a Prospective Randomized Control Trial
Brief Title: Comparison of Subtotal Stomach and Narrow Gastric Tube After Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/GCN-HDDD 2022
Record Dates: First submitted 2022-04-08; First posted 2022-04-25 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Cancer
Keywords: subtotal stomach; narrow gastric tube; anastomosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subtotal stomach (Experimental): The vessels at the anastomosis of right and left gastric arteries were separated, then the proximal haft of lesser curvature and cardia was resected using linear staplers.
  Interventions: Procedure: Narrow gastric tube
- Narrow gastric tube (Active Comparator): At the lesser curvature, the resection began at the point that was 5-cm from the pyloric, toward to the greater curvature, then the stomach was divided along 3 cm from the greater curvature using linear stapler.
  Interventions: Procedure: Narrow gastric tube

INTERVENTIONS:
Procedure: Narrow gastric tube — At the lesser curvature, the resection began at the point that was 5-cm from the pyloric, toward to the greater curvature, then the stomach was divided along 3 cm from the greater curvature using linear stapler

SUMMARY:
Currently, both the subtotal stomach and narrow gastric tube approaches are widely used for esophagogastric anastomosis after esophagectomy. Some stud- ies have concluded that the subtotal gastric conduit is superior to the wide gastric-tube approach, as it provides better protection of the submucosal vessels and can slightly increase gastric capacity.

Furthermore, blood perfusion significantly decreases after tubular gastric surgery.

DETAILED DESCRIPTION:
Stomach is the most common esophageal subtitute after a esophagectomy procedure, because it has a abundant blood supply and the need for only one anastomosis. However, cervical esophago-gastro anastomosis still has a high risk of complications, especially anastomosis leakage (11.9 - 25 % ).

There are three types of gastric subtitute: whole stomach, subtotal stomach and narrow gastric tube. While whole stomach and subtotal stomach has an advantage in the submucosal vascular network, a narrow tube is excellent elasticity and the ease with which it can be pulled up into the neck without tension, that could affect leakage rate.

On the other hand, after esophagectomy, nutrition status and quality of life (QoL) had decreased due to effect of adjuvant therapy, lower quantity of food intake, gastro-esophageal reflux and other postoperative syndromes. Several studies had shown the affect of the width of gastric tube to the postoperative nutrition and QoL, however, the results were not homogenous. This study aims to compared two types of gastric subtitute after esophagectomy: subtotal stomach and narrow gastric tube

ELIGIBILITY:
Inclusion Criteria:

* Pathologic finding by esophageal endoscopy: confirmed esophageal cancer.
* Indication for esophagectomy
* Age: 18 - 80 year old
* Tumor located at the middle or lower third of the esophagus
* ASA score: ≤ 3
* Informed consent patients (explanation about our clinical trials is provided to the patients or patrons, if patient is not available)

Exclusion Criteria:

* Concurrent cancer or patient who was treated due to other cancer before the patient was diagnosed esophageal cancer
* Pregnant patient
* Using colon or intesinal conduit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-03 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Early complications (30-day complications): rate of anastomotic leakage | 30 days after surgery
  Comparison of the rate of anastomotic leakage. All complications will be classified according to the Clavien-Dindo classification.
Early complications (30-day complications): rate of anastomotic stricture | 30 days after surgery
  Comparison of the rate of anastomotic stricture. All complications will be classified according to the Clavien-Dindo classification.
Early complications (30-day complications): rate of bleeding | 30 days after surgery
  Comparison of the rate of bleeding. All complications will be classified according to the Clavien-Dindo classification.
Early complications (30-day complications): rate of pneumonia | 30 days after surgery
  Comparison of the rate of pneumonia. All complications will be classified according to the Clavien-Dindo classification.
Early complications (30-day complications): rate of mortality. | 30 days after surgery
  Comparison of the rate of anastomotic leakage. All complications will be classified according to the Clavien-Dindo classification.
Early complications (30-day complications): rate of reoperation. | 30 days after surgery
  Comparison of the rate of reoperation. All complications will be classified according to the Clavien-Dindo classification.
Early outcomes (30-day post operative): length of hospital stay. | 30 days after surgery
  Comparison of the length of hospital stay.
Early outcomes (30-day post operative): day of oral intake. | 30 days after surgery
  Comparison of the day of oral intake.

SECONDARY OUTCOMES:
Postoperative nutritional status: body weight | 6, 12 months and 1 year after surgery
  Comparison of body weight at 6, 12 months and every year after surgery
Postoperative nutritional status: serum total protein | 6, 12 months and 1 year after surgery
  Comparison of serum total protein at 6, 12 months and every year after surgery
Postoperative nutritional status: albumin level | 6, 12 months and 1 year after surgery
  Comparison of albumin level at 6, 12 months and every year after surgery
Postoperative nutritional status: hemoglobin | 6, 12 months and 1 year after surgery
  Comparison of hemoglobin at 6, 12 months and every year after surgery
Reflux esophagitis | 6, 12 months and 1 year after surgery
  Reflux esophagitis will be evaluated using the Los Angeles classification at 6, 12 months and every year after surgery
Residue Gastritis Bile | 6, 12 months and 1 year after
  RGB (Residue Gastritis Bile) classification will be used to evaluate status of remnant stomach 6 to 12 months after surgery
Patients' health-related quality of life | 6, 12 months and 1 year after
  Patients' health-related quality of life will be evaluated using GSRS (Gastrointestinal Symptom Rating Scale) score at 6, 12 months and every year after surgery
Late complications: anastomotic stricture | 6, 12 months and 1 year after
  Comparison of the rate anastomotic stricture complications during the follow-up period
Late complications: anastomotic ulcer | 6, 12 months and 1 year after
  Comparison of anastomotic ulcer during the follow-up period
Others late complications | 6, 12 months and 1 year after
  Comparison of other late complications during the follow-up period
Oncological outcomes: overall survival rate | 6, 12 months and 1 year after
  Comparison of overall survival rate during the follow-up period
Oncological outcomes: rate of death due to the cancer | 6, 12 months and 1 year after
  Comparison of rate of death due to the cancer, and death from all causes during the follow-up period
Oncological outcomes: recurrence, metastasis | 6, 12 months and 1 year after
  Comparison of recurrence, metastasis during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Long D Vo, MD, PhD, Study Director — University Medical Center, HCMC, VN
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No